CLINICAL TRIAL: NCT00003330
Title: Phase I Clinical Trials of IV rhIL-12 With or Without a Test-Dose in Patients With Advanced Malignancies (rhIL-12 NSC# 672423)
Brief Title: Interleukin-12 in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066286; BIH-97-1083; NCI-T97-0053
Record Dates: First submitted 1999-11-01; First posted 2004-05-20 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2001-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Interleukin-12 Subunit p35

ARMS (1):
- Arm I (Experimental): See detailed description.
  Interventions: Biological: recombinant interleukin-12

INTERVENTIONS:
Biological: recombinant interleukin-12

SUMMARY:
Phase I trial to study the effectiveness of interleukin-12 in treating patients who have advanced cancer. Interleukin-12 may kill tumor cells by stopping blood flow to the tumor and by stimulating a person's white blood cells to kill cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the toxicity profile and maximum tolerated dose (MTD) of intravenous interleukin-12 (IL-12) administered biweekly for 6-18 weeks in the presence and absence of a test dose in patients with metastatic or unresectable malignancies.

II. Determine the optimal timing for administration of an IL-12 test dose, based on its impact on secondary biologic parameters in these patients.

III. Determine the antitumor effects of IL-12 administered according to this schedule, with and without a test dose, in these patients.

IV. Determine the effect of a test dose on toxicity profile, MTD, tumor response and various biologic phenomena in serum, and, where possible, tumor and liver in these patients.

OUTLINE: This is a 3-part dose escalation study.

In Part A, patients receive intravenous interleukin-12 (IL-12) twice a week for 6 weeks. Courses are repeated until patients achieve a complete response or there is disease progression. Dose escalation of IL-12 continues in cohorts of 3-6 patients until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose below that at which 2 of 6 patients experience dose limiting toxicity (DLT).

In Part B, patients receive a single test dose of IL-12 administered intravenously at a 1, 2, or 3 week interval prior to starting the multidose twice a week regimen as in Part A. Cohorts of 4 patients will receive IL-12 at the MTD obtained in Part A.

In Part C, patients receive IL-12 at one dose level above the MTD obtained in Part A using the optimal schedule for the test dose determined in Part B. Dose escalation continues in cohorts of 3-6 patients until the MTD is determined. The MTD is defined as the dose below that at which 2 of 6 patients experience DLT. Patients may continue to receive IL-12 until they have no measurable disease or until disease progression.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Advanced measurable or evaluable disease that is clearly progressive
* No brain metastases

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: ECOG 0-1 Karnofsky 80-100%
* Life expectancy: At least 3 months
* WBC greater than 4,000/mm3
* Platelet count greater than 100,000/mm3
* Bilirubin less than 1.5 mg/dL
* SGOT/SGPT less than 2 times normal
* Creatinine less than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* No congestive heart failure
* No coronary artery disease
* No serious cardiac arrhythmias
* No evidence of prior myocardial infarction on EKG
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Not HIV positive
* No seizure disorders
* No active infection that requires antibiotic therapy
* No significant medical disease other than the malignancy

PRIOR CONCURRENT THERAPY:

* No more than 2 prior biological response modifier treatment regimen
* No immunotherapy within the past 4 weeks
* No prior interleukin-12
* No more than 2 prior chemotherapy regimens
* At least 4 weeks since chemotherapy and recovered
* At least 6 weeks since nitrosoureas or mitomycin and recovered
* No concurrent chemotherapy
* At least 4 weeks since hormone therapy and recovered
* No concurrent hormone therapy
* No concurrent corticosteroids
* At least 4 weeks since radiotherapy and recovered
* No concurrent radiotherapy
* No organ allografts
* At least 2 weeks since intravenous antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 1998-07; Primary Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B. Atkins, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Gollob JA, Mier JW, Veenstra K, McDermott DF, Clancy D, Clancy M, Atkins MB. Phase I trial of twice-weekly intravenous interleukin 12 in patients with metastatic renal cell cancer or malignant melanoma: ability to maintain IFN-gamma induction is associated with clinical response. Clin Cancer Res. 2000 May;6(5):1678-92. PMID 10815886
- [Result] Gollob JA, Veenstra KG, Mier JW, Atkins MB. Agranulocytosis and hemolytic anemia in patients with renal cell cancer treated with interleukin-12. J Immunother. 2001 Jan-Feb;24(1):91-8. doi: 10.1097/00002371-200101000-00011. PMID 11211153